CLINICAL TRIAL: NCT00581035
Title: A Randomised Open Label Phase 4 Study to Evaluate the Safety and Immunogenicity of Concomitant Prevenar and Meningitec Compared to Prevenar Alone and Meningitec Alone When Used as Part of the Routine Vaccination Series in Healthy Infants
Brief Title: Study Evaluating the Safety and Ability to Produce Immune Response of Prevenar and Meningitec Given at the Same Time
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6114A1-500
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: Meningococcal disease; pneumococcal disease; meningitis
MeSH Terms: conditions — Meningococcal Infections; Pneumococcal Infections; Meningitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Prevenar and Meningitec
  Interventions: Biological: Prevenar and Meningitec
- 2 (Experimental): Prevenar
  Interventions: Biological: Prevenar
- 3 (Experimental): Meningitec
  Interventions: Biological: Meningitec

INTERVENTIONS:
Biological: Prevenar and Meningitec — 1 dose of Prevenar at 2,3.5,6 and 12 months and 1 dose of Meningitec at 2,6 and 12 months
  Arms: 1
Biological: Prevenar — 1 dose at 2,3.5,6 and 12 months
  Arms: 2
Biological: Meningitec — 1 dose at 2,6 and 12 months
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of concomitant Prevenar and Meningitec compared to Prevenar alone and Meningitec alone when used as part of the routine vaccination series in healthy infants

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 6 to 9 weeks

Ages: 42 Days to 63 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 712 (Actual)
Dates: Start 2006-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The pneumococcal and meningococcal responses achieved after the infant series | 7 months

SECONDARY OUTCOMES:
The pneumococcal and meningococcal responses achieved after the toddler dose | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer